CLINICAL TRIAL: NCT01431573
Title: Combined Wake Therapy, Light Therapy, and Lithium for Bipolar and Refractory Depression
Brief Title: Wake Therapy in the Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, David J. Hellerstein, Principal Investigator, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5491/7316R; IRB 5491 (Other Grant/Funding Number: there is no grantor or funder)
Record Dates: First submitted 2011-08-12; First posted 2011-09-09 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression | interventions — Lithium; Lithium Carbonate

STUDY DESIGN:
Masking Description: This is an "open label" study so all participants know what the treatment is.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wake Therapy + light box +/- lithium (Experimental): * Bipolar patients must take lithium; others do not take lithium
  * all patients are hospitalized for a week during which they do not sleep on alternating nights
  * for six weeks, including the week in the hospital all patients sit in front of bright lights at specified times and for specified durations
  Interventions: Behavioral: Wake Therapy; Device: light box; Drug: Lithium

INTERVENTIONS:
Behavioral: Wake Therapy — Maintaining wakefulness on alternating nights over 7 days, with continued sleep deprivation the next day.
Device: light box — use of a lightbox titrated between 15-60 minutes (typically 30 minutes), timed according to chronotype score on the Morningness-Eveningness Questionnaire
  Other Names: Day Light
Drug: Lithium — For patients not already taking lithium, dose will start at 600 mg daily (all in the evening) and be adjusted in 300 mg/d increments according to weekly blood levels (i.e., lithium dose may be changed once a week if most recent blood level is too low; if too high, it will be decreased or temporarily discontinued as clinically indicated; 150 mg increments will be utilized if multiples of 300 mg result in intolerance or blood levels outside the target range (0.6 - 1.0 mEq/L)
  Other Names: Lithobid, lithium carbonate

SUMMARY:
This pilot study seeks to replicate previous findings that sleep deprivation results in marked improvement in depression symptoms, as well as to test whether concurrent treatment with Light Therapy and Lithium are successful in locking in and maintaining therapeutic effects in both bipolar and unipolar depressed subjects.

DETAILED DESCRIPTION:
Both refractory depression and bipolar depression are difficult to treat. A night of complete sleep deprivation has been shown to result in marked improvement in 60% of depressed patients, although maintenance of therapeutic effects have not been sustained with wake therapy alone. This pilot study will assess the effectiveness of wake therapy in treating both bipolar depression (5 participants)and major depression (5 participants), as well as the effectiveness of concomitant light therapy and lithium in maintaining the therapeutic effects. Participants will undergo direct observation in the hospital for one week during initial treatment with alternating nights of sleep deprivation, light therapy and lithium treatment, and then will be seen weekly as outpatients for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. current major depressive episode (MDD, BP-I or BP-II)
2. if not BP-I or BP-II, treatment refractory to ≥ 2 adequately used antidepressants having different mechanisms
3. If BP-I or BP-II, treatment refractory to ≥ 1 standard treatment, such as lithium or valproate
4. physically healthy
5. age 18-75
6. not taking current antidepressants(antidepressants deemed effective will not be discontinued

Exclusion Criteria:

1. medically unstable condition
2. past intolerance of lithium (bipolar only)
3. history of (or current) psychosis or epilepsy
4. current (past six months) drug or alcohol abuse/dependence
5. pregnancy
6. contraindication to lithium (bipolar only)
7. significant retinal pathology (e.g., retinitis pigmentosa, macular degeneration)
8. currently taking effective antidepressant
9. cognitive dysfunction
10. Parkinson's Disease
11. Thyroid Stimulating Hormone > 5 milli International Units/Liter
12. left ventricular hypertrophy
13. symptomatic mitral valve prolapse
14. abnormal creatinine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Depression Evaluation Service - New York State Psychiatric Institute, New York, New York
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- See also: Depression Evaluation Service — http://www.depression-nyc.org
- See also: Columbia University Psychiatry — http://columbiapsychiatry.org
- See also: New York State Psychiatric Institute — http://nyspi.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Wake Therapy + Light Box +/- Lithium: * Bipolar patients must take lithium; others do not take lithium
  * all patients are hospitalized for a week during which they do not sleep on alternating nights
  * for six weeks, including the week in the hospital all patients sit in front of bright lights at specified times and for specified durations
  Wake Therapy: Maintaining wakefulness on alternating nights over 7 days, with continued sleep deprivation the next day.
  light box: use of a lightbox titrated between 15-60 minutes (typically 30 minutes), timed according to chronotype score on the Morningness-Eveningness Questionnaire
  Lithium: For patients not already taking lithium, dose will start at 600 mg daily (all in the evening) and be adjusted in 300 mg/d increments according to weekly blood levels (i.e., lithium dose may be changed once a week if most recent blood level is too low; if too high, it will be decreased or temporarily discontinued as clinically indicated; 150 mg increments will be utilized if multiples of 300 mg result in intolerance or blood levels outside the target range (0.6 - 1.0 mEq/L)
Period: Overall Study
Arm/Group | Wake Therapy + Light Box +/- Lithium
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Structured Interview for the Hamilton Depression Scale With Atypical Depression Supplement(SIGH-ADS)
Description: This is a structured interview to obtain 17 Hamilton Depression Rating Scale ratings, with 8 additional items added to measure reverse vegetative features common in bipolar depression and depression with atypical features. There are total 25 items, score ranges from 0 to 90. Higher score means worse depression.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 8
score on a scale | 16.6 (5.5)

2. Secondary Outcome: Morningness-Eveningness Questionnaire (MEQ),
Description: This is a standard self-report instrument for measuring the extent to which an individual is an "early bird" vs. a "night owl," asking a variety of questions concerning the time of day individuals prefer engagement in various activities. Scores correlate highly with biologic measures of circadian rhythm phase and will be used to custom program the timing of each patient's light therapy and habitual sleep
  Numerical scales: Multiple choice, 4-5 point scale. The sum gives a score ranging from 16 to 86; scores of 41 and below indicate "evening types", scores of 59 and above indicate "morning types", scores between 42-58 indicate "intermediate types"; 49.8% of the total population was classified as morning type compared to 5.6% having an evening-type preference
Time Frame: up to 6 weeks
Population: One patient did not complete the Week 6 assessments, mean and standard deviation are based on the 7 subjects who completed the week 6 assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 7
score on a scale | 45.3 (11.3)

3. Secondary Outcome: Symptom Check List (SCL-90)
Description: This a standard listing covering most major categories of psychiatric symptoms. It allows measurement not only of depressive symptoms over time, but also other common symptoms, such as those of panic attacks or other anxiety disorders. It consists of 90 items that yields nine scores along primary symptom dimensions and three scores among global distress indices.
  Each item scores 0-4, higher scores indicate greater distress.
  Mean of the respective item scores are used. Range from 0-4, higher value indicate greater distress.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 8
score on a scale | 1.03 (0.44)

4. Secondary Outcome: Quick Inventory of Depressive Symptoms, Self Rated (QIDS-SR 16)
Description: The responses to this question set, adapted from John Rush's Inventory of Depressive Symptoms:
  Total QIDS scores range from 0 to 27, with scores of 5 or lower indicative of no depression, scores from 6 to 10 indicating mild depression, 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 8
score on a scale | 11.5 (4.8)

5. Secondary Outcome: Hypomania Interview Guide, Current Assessment Version (HIGH-C)
Description: The HIGH-C is structured like the SIGH-ADS, and provides assessments of manic and hypomanic symptoms , in order to help identify and quantify switches and mixed states.
  All items are scored from 0 to 4, range from 0-60. An item score of "0" indicates absence of the symptom; "1" and "2" indicate incremental levels of mild presentations short of hypomania (but typical of hyperthymia); "3" indicates moderate severity, persistent and uncharacteristic for the patient, and in most cases, observable by others(as is typical of hypomania); and "4" indicates a marked or severe symptom (typical of mania). The sum of points on all items constitutes the total HIGH-R score.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 8
score on a scale | 2.0 (1.3)

6. Secondary Outcome: Clinical Global Improvement (CGI)
Description: This is a standard measure of the clinician's overall impression of how the patient is doing. It includes two measurements, one for the patient's severity of overall symptomatology, and the other for improvement since starting treatment.
  is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wake Therapy + Light Box +/- Lithium
Number analyzed (Participants) | 8
score on a scale | 3.25 (1.04)

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Wake Therapy + Light Box +/- Lithium
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT01431573/ICF_000.pdf